CLINICAL TRIAL: NCT04382898
Title: First-in-human, Dose Titration and Expansion Trial to Evaluate Safety, Immunogenicity and Preliminary Efficacy of W_pro1 (BNT112) Monotherapy and in Combination With Cemiplimab in Patients With Prostate Cancer
Brief Title: PRO-MERIT (Prostate Cancer Messenger RNA Immunotherapy)
Acronym: PRO-MERIT
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RN5609C00; 2018-004321-86 (EudraCT Number)
Record Dates: First submitted 2020-04-21; First posted 2020-05-11 (Actual); Results first posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; PRO-MERIT; Cancer vaccine; W_pro1; BioNTech SE; RNA; mCRPC; LPC; Cemiplimab; BNT112
MeSH Terms: conditions — Prostatic Neoplasms | interventions — cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part 1 (mCRPC) - dose titration (Experimental): BNT112 monotherapy
  Enrollment into this arm is completed.
  Interventions: Biological: BNT112
- Part 2 Arm 1A (mCRPC) - expansion cohort (Experimental): BNT112 in combination with cemiplimab
  Enrollment into this arm is completed.
  Interventions: Biological: BNT112; Drug: Cemiplimab
- Part 2 Arm 1B [1] (mCRPC) - expansion cohort (Experimental): BNT112 monotherapy
  Enrollment into this arm is completed.
  Interventions: Biological: BNT112
- Part 2 Arm 2 (LPC) - expansion cohort (Experimental): BNT112 in combination with cemiplimab
  Interventions: Biological: BNT112; Drug: Cemiplimab
- Part 2 Arm 3 (LPC) - expansion cohort (Experimental): BNT112 monotherapy
  Interventions: Biological: BNT112
- Part 2 Arm 1B [2] (mCRPC) - expansion cohort (Experimental): Following progression after BNT112 monotherapy, patients in Arm 1b have the option to be treated with cemiplimab monotherapy
  Enrollment into this arm is completed.
  Interventions: Drug: Cemiplimab

INTERVENTIONS:
Biological: BNT112 — Intravenous bolus injection
  Arms: Part 1 (mCRPC) - dose titration; Part 2 Arm 1A (mCRPC) - expansion cohort; Part 2 Arm 1B [1] (mCRPC) - expansion cohort; Part 2 Arm 2 (LPC) - expansion cohort; Part 2 Arm 3 (LPC) - expansion cohort
Drug: Cemiplimab — Intravenous infusion
  Arms: Part 2 Arm 1A (mCRPC) - expansion cohort; Part 2 Arm 1B [2] (mCRPC) - expansion cohort; Part 2 Arm 2 (LPC) - expansion cohort

SUMMARY:
Open-label, multicenter, dose titration and four-arm expansion trial to evaluate the safety, tolerability, immunogenicity, and preliminary efficacy of BNT112 cancer vaccine (BNT112) monotherapy or in combination with cemiplimab in patients with metastatic castration resistant prostate cancer (mCRPC: Part 1 and Part 2 Arms 1A and 1B) and in patients with high-risk, localized prostate cancer (LPC).

As of February 2023, the trial only recruited LPC patients and no longer mCRPC patients.

DETAILED DESCRIPTION:
* BNT112 consisted of messenger ribonucleic acid (mRNA [or RNA]) targeting 5 antigens expressed in de novo and metastatic prostate cancer that were separately complexed with liposomes to form serum-stable RNA lipoplexes (RNA-LPX).
* The RNA molecules were immune-pharmacologically optimized for high stability, translational efficiency and presentation on major histocompatibility complex (MHC) class I and II molecules. The vaccine was intended for intravenous (IV) bolus injection.
* The RNA-LPX cancer vaccine induced activation of both the adaptive immune system (vaccine antigen-specific CD8+/CD4+ T cell) as well as the innate immune system (TLR7 agonism of single-stranded RNA). The physiology of efficient induction, expansion and differentiation of antigen-specific T cells was associated with programmed death receptor-1 (PD-1) upregulation on these T cells. Thus, the cancer vaccine was expected to have a synergistic mechanism of action with anti-PD-1.
* The step-up dose titration approach allowed for optimal dose management on an individual basis and accounted for inter- and intra-individual variability of the immune system.
* In summary, the mechanism of action of BNT112 both in monotherapy and in combination with anti-PD-1 immune checkpoint inhibitor cemiplimab, together with carefully selected and refined clinical setting presented a unique opportunity for patients with different stages of prostate cancer.

ELIGIBILITY:
Inclusion criteria:

* Patients were male and aged >=18 years.
* Patients had histologically confirmed prostate adenocarcinoma.
* Patients had an Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of 0 or 1.

Specific key inclusion criteria for mCRPC patients (Part 1 and Part 2 Arms 1A and 1B) - Recruitment of mCRPC patients now completed:

* Patients had histologically confirmed mCRPC and had progressed after at least 2 but no more than 3 lines of life-prolonging systemic therapy (e.g., abiraterone or enzalutamide, docetaxel, cabazitaxel) or cannot tolerate or refused any of these therapies. These lines of therapy included life-prolonging therapies administered in the metastatic hormone-sensitive setting.
* Prior surgical or chemical castration with a serum testosterone <1.7 nmol/L (50 ng/dL). If the method of castration was luteinizing hormone-releasing hormone analogue (LHRHa), there was a plan to maintain effective LHRHa therapy for the duration of the trial.
* Patients had documented mCRPC progression within 6 months prior to screening (assuming no subsequent change in treatments), as determined by the investigator.
* Patients agreed to provide an archival pre-treatment formalin-fixed, paraffin-embedded tumor sample if available.

Specific key inclusion criteria for newly diagnosed LPC patients (Part 2 Arms 2 and 3):

* Treatment-naïve patients with LPC (i.e., N0, M0). According to risk levels of the European Association of Urology Guidelines on Prostate Cancer (2018), and in line with the U.S. National Comprehensive Cancer Network (NCCN 2020), patients had at least 1 of the following:

  1. PSA >20 ng/mL or
  2. Gleason Score >7 or
  3. Localized stage >=cT2c, N0, M0 according to tumor, node, metastasis classification.
* Patients who intend to have and were suitable for a radical prostatectomy.
* Patients agreed to provide tumor sample(s) from pre-treatment diagnostic biopsy and planned post-treatment surgery.

Main exclusion criteria for all patients:

Medical conditions

* Patients with uncontrolled intercurrent illness.
* Patients with a known history or current malignancy other than the inclusion diagnosis. Note: Exceptions were patients with malignancies with a negligible risk of metastasis or death, that had been adequately treated, such as non-invasive basal cell or non-invasive squamous cell skin carcinoma, non-invasive, superficial bladder cancer, and any cancer with a complete response (CR) that lasted more than 2 years might be included.
* Patients who had major surgery (e.g., requiring general anesthesia) within 4 weeks before screening, or have not fully recovered from surgery, or had a surgery planned during the time of trial participation, except for the radical prostatectomy planned for patients in Part 2 Arms 2 and 3.
* Patients who had a known history of any of the following:

  1. Human immunodeficiency virus (HIV) 1 or 2
  2. Hepatitis B (carrier or active infection)
  3. Hepatitis C (unless considered cured 5 years post curative anti-viral therapy)
* Patients who have received or currently receive the following therapy/treatment:

  1. Chronic systemic immunosuppressive corticosteroid treatment (prednisone >5 mg daily orally [PO] or IV, or equivalent) during the trial. Note: Replacement therapy (e.g., physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is permitted.
  2. Prior treatment with other immune modulating agents that was (a) within fewer than 4 weeks (28 days) or 5 half-lives (whichever is longer) prior to the first dose of cemiplimab, or (b) associated with immune-mediated AEs that were Grade >=1 within 90 days prior to the first dose of cemiplimab, or (c) associated with toxicity that resulted in discontinuation of the immune-modulating agent.
  3. Prior treatment with other immune modulating agents for any non-cancer disease within 4 weeks or 5 half-lives of the agent (whichever is longer) before the first dose of IMP.
  4. Prior treatment with live-attenuated vaccines within 4 weeks before the first dose of IMP and during treatment with IMP.
  5. Prior treatment with an investigational drug (including investigational vaccines) within 4 weeks or 5 half-lives of the agent (whichever is longer) before the planned first dose of IMP.
  6. Therapeutic PO or IV antibiotics within 14 days prior to enrollment. Note: Patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or chronic obstructive pulmonary disease) might be enrolled.
  7. Concurrent use of herbal products that might decrease PSA levels (e.g., saw palmetto).

Specific key exclusion criteria for mCRPC Patients (Part 1 and Part 2 Arms 1A and 1B) - Recruitment of mCRPC patients now completed:

Excluded medical conditions

* Patients with toxicities from previous anti-cancer therapies that have not resolved to baseline levels or to Grade <=1 according to National Cancer Institute (NCI) CTCAE v5.0 with the exception of alopecia, anorexia, vitiligo, fatigue, hyperthyroidism, hypothyroidism, and peripheral neuropathy. Anorexia, hyperthyroidism, hypothyroidism, and peripheral neuropathy must have recovered to Grade <=2.
* Patients with clinically active brain metastases.

  1. Patients with a history of symptomatic metastatic brain or meningeal tumors might be included, if the end of definitive therapy was >3 months before the first dose of BNT112 and the patients had no clinical or radiological evidence of tumor growth.
  2. Patients with brain metastases must not be undergoing acute or chronic corticosteroid therapy or steroid taper.
  3. Patients with central nervous system symptoms should undergo a computed tomography (CT) scan or magnetic resonance imaging (MRI) of the brain to exclude new or progressive brain metastases. Spinal cord metastasis is acceptable. However, patients with spinal cord compression should be excluded.

Excluded prior or concomitant anti-cancer therapies

* Patients who received or currently receive the following anti-cancer therapy/agent:

  1. Prior radiation therapy with curative intent within 14 days before the first dose of IMP. Note: Palliative radiotherapy is allowed.
  2. Prior treatment with an anti-cancer agent (within 4 weeks or for systemic therapies after at least 5 half-lives of the drug [whichever is longer] before the first dose of IMP). Note: Prior treatment with bone resorptive therapy, such as bisphosphonates (e.g., pamidronate, zoledronic acid, etc.) and denosumab, is allowed assuming that the patients have been on stable doses for >=4 weeks prior to first dose of trial treatment.
  3. Prior treatment with anti-cancer immunomodulating agents, such as blockers of programmed death receptor-1 PD-1, programmed cell death 1 ligand 1 (PD-L1), tumor necrosis factor receptor superfamily member 9 (TNRSF9, 4-1BB, CD137), OX-40, therapeutic vaccines, cytokine treatments, or any investigational agent within 4 weeks or 5 half-lives (whichever was longer) before the first dose of IMP.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2024-01-23 (Actual); Study Completion 2024-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: BioNTech Responsible Person, Study Director — BioNTech SE
Locations (22):
- United States (5):
  - The University of Arizona Cancer Center, Tucson, Arizona
  - University of Miami Hospital & Clinics /Sylvester Comprehensive Cancer Center, Miami, Florida
  - University of Pittsburgh Cancer Inst., Pittsburgh, Pennsylvania
  - Urology San Antonio P.A., San Antonio, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
- Germany (6):
  - Universitätsklinikum Bonn, Bonn
  - Klinikum der Johann Wolfgang Goethe-Universität, Frankfurt
  - Universitätsklinikum Münster, Münster
  - Studienpraxis Urologie, Nürtingen
  - Urologische Klinik Planegg, Planegg
  - Universitätsklinikum Tübingen, Tübingen
- Hungary (5):
  - Magyar Honvédség Egészségügyi Központ (MH EK Honvédkórház), Budapest
  - Semmelweis Egyetem, Belgyógyászati Klinika, Budapest
  - Onkológiai Klinika, Debrecen
  - Szabolcs-Szatmár-Bereg Megyei Kórházak és Egyetemi Oktatókórház, Nyíregyháza
  - Szent Borbála Kórház, Tatabánya
- United Kingdom (6):
  - Cancer Research UK Cambridge Centre, Cambridge
  - Velindre Cancer Centre (VCC), Cardiff
  - University of Glasgow, Beatson WoS Cancer Centre, Glasgow
  - University College London Hospitals, London
  - The Royal Marsden Hospital, London
  - University Hospital Southampton - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial consisted of 2 parts: Part 1 (dose titration) and Part 2 (dose expansion; consisted of four arms).
Pre-assignment Details: Part 1 and Part 2 (Arms 1A and 1B) enrolled participants with metastatic castration-resistant prostate cancer (mCRPC). Part 2: Arms 2 and 3 enrolled participants with newly diagnosed high-risk localized prostate cancer (LPC). A total of 75 participants (9 participants in Part 1 and 66 in Part 2) were enrolled in this study. All participants in Part 1 and Part 2 received the same dose of cemiplimab.
Groups:
- Part 1 (mCRPC): BNT112: Participants with mCRPC received intravenous (IV) administration of BNT112 (cumulative doses ranged from 100 to 1175 micrograms [mcg]) on Days 1, 8 and 15 of Cycle 1 and Cycle 2, thereafter every 3 weeks (Q3W) starting with Day 1 of Cycle 3 for each of the 21-days treatment cycles until unacceptable toxicity or disease progression.
- Part 2 (mCRPC): Arm 1a: BNT112 + Cemiplimab: Participants with mCRPC received IV administration of BNT112 (cumulative doses ranged from 25 to 1675 mcg) on Days 1, 8 and 15 of Cycle 1 and Cycle 2, thereafter Q3W starting with Day 1 of Cycle 3 along with cemiplimab IV Q3W for each of the 21-days treatment cycles until unacceptable toxicity or disease progression.
- Part 2 (mCRPC): Arm 1b: BNT112: Participants with mCRPC received IV administration of BNT112 (cumulative doses ranged from 25 to 3575 mcg) on Days 1, 8 and 15 of Cycle 1 and Cycle 2, thereafter Q3W starting with Day 1 of Cycle 3 for each of the 21-days treatment cycles until unacceptable toxicity or disease progression.
- Part 2 (LPC): Arm 2: BNT112 + Cemiplimab: Participants with high-risk, localized prostate cancer (LPC) received IV administration of BNT112 (cumulative doses ranged from 1075 to 1075 mcg) on Days 1, 8 and 15 of Cycle 1 and Cycle 2, thereafter Q3W starting with Day 1 of Cycle 3 Q3W along with cemiplimab IV Q3W for each of the 21-days treatment cycles until unacceptable toxicity or disease progression, or up to Cycle 8 followed by radical prostatectomy.
- Part 2 (LPC): Arm 3: BNT112: Participants with high-risk LPC received IV administration of BNT112 (cumulative doses ranged from 975 to 1075 mcg) on Days 1, 8 and 15 of Cycle 1 and Cycle 2, thereafter Q3W starting with Day 1 of Cycle 3 for each of the 21-days treatment cycles until unacceptable toxicity or disease progression, or up to Cycle 8 followed by radical prostatectomy.
Period: Part 1: Dose Titration
Arm/Group | Part 1 (mCRPC): BNT112 | Part 2 (mCRPC): Arm 1a: BNT112 + Cemiplimab | Part 2 (mCRPC): Arm 1b: BNT112 | Part 2 (LPC): Arm 2: BNT112 + Cemiplimab | Part 2 (LPC): Arm 3: BNT112
Started | 9 | 0 (Part 1 and Part 2 were separate populations.) | 0 | 0 | 0
Completed | 2 | 0 | 0 | 0 | 0
Not Completed | 7 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0
Not completed — Death | 6 | 0 | 0 | 0 | 0
Period: Part 2: Dose Expansion
Arm/Group | Part 1 (mCRPC): BNT112 | Part 2 (mCRPC): Arm 1a: BNT112 + Cemiplimab | Part 2 (mCRPC): Arm 1b: BNT112 | Part 2 (LPC): Arm 2: BNT112 + Cemiplimab | Part 2 (LPC): Arm 3: BNT112
Started | 0 | 28 (Part 1 and Part 2 were separate populations.) | 27 (Part 1 and Part 2 were separate populations.) | 5 (Part 1 and Part 2 were separate populations.) | 6 (Part 1 and Part 2 were separate populations.)
Completed | 0 | 10 | 9 | 4 | 5
Not Completed | 0 | 18 | 18 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0
Not completed — Death | 0 | 17 | 13 | 1 | 0
Not completed — Progressive Disease | 0 | 0 | 1 | 0 | 0
Not completed — Study Terminated By Sponsor | 0 | 1 | 1 | 0 | 1
Not completed — Other | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on Intent to Treat (ITT) population that included all participants who were randomized to the investigational medicinal product (IMP).
Groups:
- Part 1 (mCRPC): BNT112: Participants with mCRPC received IV administration of BNT112 (cumulative doses ranged from 100 to 1175 mcg) on Days 1, 8 and 15 of Cycle 1 and Cycle 2, thereafter Q3W starting with Day 1 of Cycle 3 for each of the 21-days treatment cycles until unacceptable toxicity or disease progression.
- Part 2 (LPC): Arm 2: BNT112 + Cemiplimab: Participants with high-risk LPC received IV administration of BNT112 (cumulative doses ranged from 1075 to 1075 mcg) on Days 1, 8 and 15 of Cycle 1 and Cycle 2, thereafter Q3W starting with Day 1 of Cycle 3 along with cemiplimab IV Q3W for each of the 21-days treatment cycles until unacceptable toxicity or disease progression, or up to Cycle 8 followed by radical prostatectomy.
- Total: Total of all reporting groups
Arm/Group | Part 1 (mCRPC): BNT112 | Part 2 (mCRPC): Arm 1a: BNT112 + Cemiplimab | Part 2 (mCRPC): Arm 1b: BNT112 | Part 2 (LPC): Arm 2: BNT112 + Cemiplimab | Part 2 (LPC): Arm 3: BNT112 | Total
Number analyzed (Participants) | 9 | 28 | 27 | 5 | 6 | 75
Age, Customized [Count of Participants; unit: Participants]
  < 50 years | 0 | 0 | 0 | 0 | 0 | 0
  >= 50 - < 65 years | 1 | 7 | 11 | 3 | 4 | 26
  >= 65 - < 85 years | 8 | 20 | 16 | 2 | 2 | 48
  >= 85 years | 0 | 1 | 0 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 9 | 28 | 27 | 5 | 6 | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 4 | 0 | 0 | 0 | 4
  Not Hispanic or Latino | 9 | 23 | 27 | 4 | 6 | 69
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 2 | 1 | 5
  White | 8 | 27 | 26 | 3 | 5 | 69
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLT criteria were defined as following: any treatment-emergent adverse events (TEAE) of Grade 5 intensity; hematological toxicities (Grade 3 and 4 febrile neutropenia, Grade 4 thrombocytopenia, Grade 3 and 4 hemorrhage associated with thrombocytopenia of Grade greater than or equal to [>=] 3, Grade 4 anemia); and non-hematological toxicities (Grade 4 cytokine release syndrome [CRS], Grade 3 CRS which has not improved to Grade 1 or resolved within 48 hours; any Grade >=3 non-hematological TEAE at least possibly related which occurs during the first BNT112 cancer vaccine treatment cycle).
Time Frame: Cycle 1 (21 days)
Population: Analysis was performed on the DLT evaluation set that included all participants who received IMP and completed the DLT evaluation period and met the minimum exposure criterion or experienced a DLT during Cycle 1. Data for this outcome measure was not planned to be collected and analyzed for Part 2 arms.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 (mCRPC): BNT112
Number analyzed (Participants) | 9
Participants | 2

2. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs and TEAEs Related to Trial Procedure
Description: TEAE: any adverse event (AE) with an onset date on or after the first administration of investigational medicinal product (IMP) or worsened after first administration of IMP. AEs with an onset date more than 30 days after last dose of BNT112 or 90 days after last dose of cemiplimab (for Part 2, Arm 1a and Arm 2) were only considered as TEAEs if assessed as related to IMP by the investigator. Serious adverse event (SAE): any untoward medical occurrence that, at any dose: resulted in death; was life-threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent disability/incapacity; was a congenital anomaly/birth defect or was another medically important condition. AEs were graded for severity using National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0 (NCI-CTCAE v5.0), where Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe; Grade 4 - Life-threatening consequences; Grade 5: Death related to AE.
Time Frame: From Baseline up to 30 days after the last dose of BNT112 (for Part 1 and Part 2 Arms 1b and 3) or up to 90 days after the last dose of cemiplimab (for Part 2, Arm 1a and Arm 2) (up to 4 years and 1 month)
Population: Analysis was performed on safety set that included all participants who received at least 1 dose of the IMP.
Measure: Count of Participants; unit: Participants
Groups:
- Part 2 (LPC): Arm 2: BNT112 + Cemiplimab: Participants with high-risk LPC received IV administration of BNT112 (cumulative doses ranged from 1075 to 1075 mcg) on Days 1, 8 and 15 of Cycle 1 and Cycle 2, thereafter Q3W starting with Day 1 of Cycle 3 Q3W along with cemiplimab IV Q3W for each of the 21-days treatment cycles until unacceptable toxicity or disease progression, or up to Cycle 8 followed by radical prostatectomy.
Arm/Group | Part 1 (mCRPC): BNT112 | Part 2 (mCRPC): Arm 1a: BNT112 + Cemiplimab | Part 2 (mCRPC): Arm 1b: BNT112 | Part 2 (LPC): Arm 2: BNT112 + Cemiplimab | Part 2 (LPC): Arm 3: BNT112
Number analyzed (Participants) | 9 | 28 | 27 | 5 | 6
Participants
  TEAEs | 8 | 28 | 26 | 5 | 6
  Serious TEAE | 5 | 5 | 9 | 2 | 2
  Grade >= 3 TEAEs | 7 | 15 | 15 | 1 | 4
  Grade 5 TEAEs | 2 | 0 | 1 | 0 | 0
  TEAEs related to trial procedure | 1 | 1 | 0 | 1 | 2

3. Primary Outcome: Part 2 Arm 1a: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants with a complete response (CR) or partial response (PR) as per Prostate Cancer Working Group 3 (PCWG3) criteria as determined by the investigator. Participants not meeting the criteria for CR or PR, including those without any post-baseline tumor assessments, were considered as non-responders. CR was defined as the disappearance of all target lesions, with a reduction in short axis to <10 mm in any pathological lymph nodes and no new lesions. PR was defined as 30% decrease in the sum of the longest diameter of target lesions.
Time Frame: From start of treatment up to 46 weeks
Population: Analysis was performed on modified Intent to Treat population (mITT) population that included all participants who were randomized to the IMP and had a baseline and at least one post-baseline (i.e., one on-treatment or post-treatment) tumor assessment (clinical or imaging assessment). Data for this outcome measure was not planned to be collected and analyzed for Part 2: Arms 2 and 3.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2 (mCRPC): Arm 1a: BNT112 + Cemiplimab
Number analyzed (Participants) | 27
percentage of participants | 0 [0.0 to 12.8]
Statistical Analysis 1: Comparison: Part 2 (mCRPC): Arm 1a: BNT112 + Cemiplimab; Test type: Superiority; p = 0.1041, Fisher Exact

4. Secondary Outcome: Number of Participants Reporting Change From Baseline in Prostate-specific Antigen (PSA) Levels
Description: Participants blood samples were tested for levels of PSA to track the progression of prostate cancer. PSA decline categories of No decline, 0 to 25%, >25% to 50%, and >50% compared to baseline during treatment according to PCWG3 (as reported by the investigator) are reported in this outcome measure. EOT in the timeframe below refers to End of treatment.
Time Frame: Day8 (Cycles1&2 only), Day1 Cycle 2 & Day 15 (Cycles1,2 & 8 only) (each cycle of 21-days), & EOT (30 days after last dose of BNT112 [Part 1 & Part 2 Arms 1b & 3] or 90 days after last dose of cemiplimab [Part 2, Arm 1a & Arm 2] [up to 4 years & 1 months])
Population: Analysis was performed on mITT population. Here, "Overall number of participants analyzed" = participants with available data for this outcome measure and number analyzed signifies participants with available data for each specified category at respective visit and "0" in the number analyzed field signifies that no participants were available for analysis at the specified visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 (mCRPC): BNT112 | Part 2 (mCRPC): Arm 1a: BNT112 + Cemiplimab | Part 2 (mCRPC): Arm 1b: BNT112 | Part 2 (LPC): Arm 2: BNT112 + Cemiplimab | Part 2 (LPC): Arm 3: BNT112
Number analyzed (Participants) | 8 | 24 | 23 | 5 | 6
Participants
  Cycle 1 Day 8: No decline: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1
  Cycle 1 Day 8: No decline |  |  |  |  | 1
  Cycle 1 Day 8: 0 to 25%: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1
  Cycle 1 Day 8: 0 to 25% |  |  |  |  | 0
  Cycle 1 Day 8: Greater than (>) 25% to 50%: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1
  Cycle 1 Day 8: Greater than (>) 25% to 50% |  |  |  |  | 0
  Cycle 1 Day 8: >50%: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1
  Cycle 1 Day 8: >50% |  |  |  |  | 0
  Cycle 1 Day 15: No decline: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1
  Cycle 1 Day 15: No decline |  |  |  |  | 0
  Cycle 1 Day 15: 0 to 25%: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1
  Cycle 1 Day 15: 0 to 25% |  |  |  |  | 0
  Cycle 1 Day 15: >25% to 50%: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1
  Cycle 1 Day 15: >25% to 50% |  |  |  |  | 1
  Cycle 1 Day 15: >50%: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1
  Cycle 1 Day 15: >50% |  |  |  |  | 0
  Cycle 2 Day 1: No decline | 6 | 21 | 19 | 1 | 0
  Cycle 2 Day 1: 0 to 25% | 2 | 3 | 2 | 1 | 1
  Cycle 2 Day 1: Greater than (>) 25% to 50% | 0 | 0 | 1 | 0 | 1
  Cycle 2 Day 1: >50% | 0 | 0 | 1 | 3 | 4
  Cycle 2 Day 8: No decline: number analyzed (Participants) | 1 | 0 | 0 | 0 | 1
  Cycle 2 Day 8: No decline | 1 |  |  |  | 0
  Cycle 2 Day 8: 0 to 25%: number analyzed (Participants) | 1 | 0 | 0 | 0 | 1
  Cycle 2 Day 8: 0 to 25% | 0 |  |  |  | 0
  Cycle 2 Day 8: > 25% to 50%: number analyzed (Participants) | 1 | 0 | 0 | 0 | 1
  Cycle 2 Day 8: > 25% to 50% | 0 |  |  |  | 0
  Cycle 2 Day 8: >50%: number analyzed (Participants) | 1 | 0 | 0 | 0 | 1
  Cycle 2 Day 8: >50% | 0 |  |  |  | 1
  Cycle 2 Day 15: No decline: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1
  Cycle 2 Day 15: No decline |  |  |  |  | 0
  Cycle 2 Day 15: 0 to 25%: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1
  Cycle 2 Day 15: 0 to 25% |  |  |  |  | 0
  Cycle 2 Day 15: > 25% to 50%: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1
  Cycle 2 Day 15: > 25% to 50% |  |  |  |  | 0
  Cycle 2 Day 15: >50%: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1
  Cycle 2 Day 15: >50% |  |  |  |  | 1
  Cycle 8 Day 15: No decline: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0
  Cycle 8 Day 15: No decline |  |  | 1 |  |
  Cycle 8 Day 15: 0 to 25%: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0
  Cycle 8 Day 15: 0 to 25% |  |  | 0 |  |
  Cycle 8 Day 15: > 25% to 50%: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0
  Cycle 8 Day 15: > 25% to 50% |  |  | 0 |  |
  Cycle 8 Day 15: >50%: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0
  Cycle 8 Day 15: >50% |  |  | 0 |  |
  EOT: No decline: number analyzed (Participants) | 7 | 19 | 19 | 4 | 3
  EOT: No decline | 7 | 17 | 19 | 0 | 0
  EOT: 0 to 25%: number analyzed (Participants) | 7 | 19 | 19 | 4 | 3
  EOT: 0 to 25% | 0 | 2 | 0 | 0 | 0
  EOT: > 25% to 50%: number analyzed (Participants) | 7 | 19 | 19 | 4 | 3
  EOT: > 25% to 50% | 0 | 0 | 0 | 0 | 0
  EOT: >50%: number analyzed (Participants) | 7 | 19 | 19 | 4 | 3
  EOT: >50% | 0 | 0 | 0 | 4 | 3

5. Secondary Outcome: Number of Participants Reporting Change From Baseline in PSA Doubling Time (PSADT)
Description: Participants blood samples were tested for levels of PSA to track the progression of prostate cancer. PSADT was calculated using a linear regression model of the natural logarithm of PSA values and time. PSA doubling time compared to baseline during the treatment period for the following categories: 0 - 3 months; >3 - 6 months; >6 - 9 months; >9 - 12 months; >12 - 18 months; >18 - 24 months; >24 months and declining are reported in this outcome measure.
Time Frame: Cycle 4 Day 1, Cycle 8 Day 1, Cycle 12 Day 1 (each cycle duration=21 days)
Population: Analysis was performed on mITT population. Here, "Overall number of participants analyzed" = participants with available data for this outcome measure and number analyzed signifies participants with available data for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 (mCRPC): BNT112 | Part 2 (mCRPC): Arm 1a: BNT112 + Cemiplimab | Part 2 (mCRPC): Arm 1b: BNT112 | Part 2 (LPC): Arm 2: BNT112 + Cemiplimab | Part 2 (LPC): Arm 3: BNT112
Number analyzed (Participants) | 6 | 21 | 19 | 5 | 6
Participants
  Cycle 4 Day 1: 0 - 3 months: number analyzed (Participants) | 6 | 21 | 19 | 5 | 5
  Cycle 4 Day 1: 0 - 3 months | 5 | 16 | 11 | 1 | 0
  Cycle 4 Day 1: >3 - 6 months: number analyzed (Participants) | 6 | 21 | 19 | 5 | 5
  Cycle 4 Day 1: >3 - 6 months | 0 | 2 | 2 | 0 | 0
  Cycle 4 Day 1: >6 - 9 months: number analyzed (Participants) | 6 | 21 | 19 | 5 | 5
  Cycle 4 Day 1: >6 - 9 months | 1 | 1 | 2 | 0 | 0
  Cycle 4 Day 1: >9 - 12 months: number analyzed (Participants) | 6 | 21 | 19 | 5 | 5
  Cycle 4 Day 1: >9 - 12 months | 0 | 0 | 0 | 0 | 0
  Cycle 4 Day 1: >12 - 18 months: number analyzed (Participants) | 6 | 21 | 19 | 5 | 5
  Cycle 4 Day 1: >12 - 18 months | 0 | 0 | 0 | 0 | 0
  Cycle 4 Day 1: >18 - 24 months: number analyzed (Participants) | 6 | 21 | 19 | 5 | 5
  Cycle 4 Day 1: >18 - 24 months | 0 | 0 | 1 | 0 | 0
  Cycle 4 Day 1: >24 months: number analyzed (Participants) | 6 | 21 | 19 | 5 | 5
  Cycle 4 Day 1: >24 months | 0 | 0 | 0 | 0 | 0
  Cycle 4 Day 1: Declining: number analyzed (Participants) | 6 | 21 | 19 | 5 | 5
  Cycle 4 Day 1: Declining | 0 | 2 | 3 | 4 | 5
  Cycle 8 Day 1: 0 - 3 months: number analyzed (Participants) | 4 | 13 | 15 | 5 | 6
  Cycle 8 Day 1: 0 - 3 months | 3 | 6 | 8 | 0 | 0
  Cycle 8 Day 1: >3 - 6 months: number analyzed (Participants) | 4 | 13 | 15 | 5 | 6
  Cycle 8 Day 1: >3 - 6 months | 0 | 5 | 1 | 0 | 0
  Cycle 8 Day 1: >6 - 9 months: number analyzed (Participants) | 4 | 13 | 15 | 5 | 6
  Cycle 8 Day 1: >6 - 9 months | 0 | 1 | 0 | 0 | 0
  Cycle 8 Day 1: >9 - 12 months: number analyzed (Participants) | 4 | 13 | 15 | 5 | 6
  Cycle 8 Day 1: >9 - 12 months | 0 | 0 | 2 | 0 | 0
  Cycle 8 Day 1: >12 - 18 months: number analyzed (Participants) | 4 | 13 | 15 | 5 | 6
  Cycle 8 Day 1: >12 - 18 months | 0 | 0 | 1 | 0 | 0
  Cycle 8 Day 1: >18 - 24 months: number analyzed (Participants) | 4 | 13 | 15 | 5 | 6
  Cycle 8 Day 1: >18 - 24 months | 0 | 0 | 0 | 0 | 0
  Cycle 8 Day 1: > 24 months: number analyzed (Participants) | 4 | 13 | 15 | 5 | 6
  Cycle 8 Day 1: > 24 months | 1 | 0 | 1 | 0 | 0
  Cycle 8 Day 1: Declining: number analyzed (Participants) | 4 | 13 | 15 | 5 | 6
  Cycle 8 Day 1: Declining | 0 | 1 | 2 | 5 | 6
  Cycle 12 Day 1: 0 - 3 months: number analyzed (Participants) | 3 | 7 | 6 | 4 | 3
  Cycle 12 Day 1: 0 - 3 months | 3 | 2 | 0 | 0 | 0
  Cycle 12 Day 1: >3 - 6 months: number analyzed (Participants) | 3 | 7 | 6 | 4 | 3
  Cycle 12 Day 1: >3 - 6 months | 0 | 3 | 1 | 0 | 0
  Cycle 12 Day 1: >6 - 9 months: number analyzed (Participants) | 3 | 7 | 6 | 4 | 3
  Cycle 12 Day 1: >6 - 9 months | 0 | 1 | 2 | 0 | 0
  Cycle 12 Day 1: >9 - 12 months: number analyzed (Participants) | 3 | 7 | 6 | 4 | 3
  Cycle 12 Day 1: >9 - 12 months | 0 | 0 | 1 | 0 | 0
  Cycle 12 Day 1: >12 - 18 months: number analyzed (Participants) | 3 | 7 | 6 | 4 | 3
  Cycle 12 Day 1: >12 - 18 months | 0 | 0 | 0 | 0 | 0
  Cycle 12 Day 1: >18 - 24 months: number analyzed (Participants) | 3 | 7 | 6 | 4 | 3
  Cycle 12 Day 1: >18 - 24 months | 0 | 0 | 0 | 0 | 0
  Cycle 12 Day 1: > 24 months: number analyzed (Participants) | 3 | 7 | 6 | 4 | 3
  Cycle 12 Day 1: > 24 months | 0 | 0 | 0 | 0 | 0
  Cycle 12 Day 1: Declining: number analyzed (Participants) | 3 | 7 | 6 | 4 | 3
  Cycle 12 Day 1: Declining | 0 | 1 | 2 | 4 | 3

6. Secondary Outcome: Number of Participants With PSA Decline of >=50%
Description: Participants blood samples were tested for levels of PSA to track the progression of prostate cancer. Participants with PSA decline of >=50% compared to baseline according to PCWG3 (as reported by the investigator) are reported in this outcome measure. EOT in the timeframe below refers to End of treatment.
Time Frame: as for outcome 4
Population: Analysis was performed on mITT population. Here, "Overall number of participants analyzed" = participants with available data for this outcome measure and "number analyzed" signifies participants with available data for each specified category at respective visit and "0" in the number analyzed field signifies that no participants were available for analysis at the specified visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 (mCRPC): BNT112 | Part 2 (mCRPC): Arm 1a: BNT112 + Cemiplimab | Part 2 (mCRPC): Arm 1b: BNT112 | Part 2 (LPC): Arm 2: BNT112 + Cemiplimab | Part 2 (LPC): Arm 3: BNT112
Number analyzed (Participants) | 8 | 24 | 23 | 5 | 6
Participants
  Cycle 1 Day 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1
  Cycle 1 Day 8 |  |  |  |  | 0
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1
  Cycle 1 Day 15 |  |  |  |  | 0
  Cycle 2 Day 1 | 0 | 0 | 1 | 3 | 4
  Cycle 2 Day 8: number analyzed (Participants) | 1 | 0 | 0 | 0 | 1
  Cycle 2 Day 8 | 0 |  |  |  | 1
  Cycle 2 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1
  Cycle 2 Day 15 |  |  |  |  | 1
  Cycle 8 Day 15: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0
  Cycle 8 Day 15 |  |  | 0 |  |
  EOT: number analyzed (Participants) | 7 | 19 | 19 | 4 | 3
  EOT | 0 | 0 | 0 | 4 | 3

7. Secondary Outcome: Part 1: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants with a CR or PR as per PCWG3 criteria as determined by the investigator. Participants not meeting the criteria for CR or PR, including those without any post-baseline tumor assessments, were considered as non-responders. CR was defined as the disappearance of all target lesions, with a reduction in short axis to <10 mm in any pathological lymph nodes and no new lesions. PR was defined as 30% decrease in the sum of the longest diameter of target lesions.
Time Frame: From start of treatment up to 27 weeks
Population: Analysis was performed on mITT population. Data for this outcome measure was not planned to be collected and analyzed for Part 2: Arms 2 and 3.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1 (mCRPC): BNT112
Number analyzed (Participants) | 9
percentage of participants | 0 [0.0 to 33.6]

8. Secondary Outcome: Part 2: Arms 2 and 3: Number of Participants With Tumor Response Post-Treatment
Description: The best overall response was defined as a single best response status at any tumor response assessment after first administration of IMP and prior to or at the start date of the first subsequent anti-cancer therapy. Overall response of progressive disease within 14 days after the start date of first subsequent anti-cancer therapy was considered. The following order of tumor response categories were used, where "Complete Response" is the best category: Complete Response (CR) - Partial Response (PR) - Stable Disease (SD) - Progressive Disease (PD) - Not Evaluable (NE) - Missing. CR: disappearance of all target lesions, with reduction in short axis to <10 mm in any pathological lymph nodes and no new lesions. PR:30% decrease in the sum of the longest diameter of target lesions. PD: progression of target lesions (sum of diameter increase to nadir of >=20% and by >=5 mm), progression of existing non-target lesions, or appearance of 1 or more new lesions.SD: no evidence of PD, CR or PR.
Time Frame: From start of treatment up to 25 weeks (Arm 2) and up to 26 weeks (Arm 3)
Population: Analysis was performed on mITT population. Data for this outcome measure was not planned to be collected and analyzed for Part 1 and Part 2: Arms 1a and 1b.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 (LPC): Arm 2: BNT112 + Cemiplimab | Part 2 (LPC): Arm 3: BNT112
Number analyzed (Participants) | 5 | 6
Participants
  Complete Response (CR) | 0 | 0
  Partial Response (PR) | 3 | 3
  Stable Disease (SD) | 2 | 2
  Progressive Disease (PD) | 0 | 0
  Not Evaluable (NE) | 0 | 0
  Missing | 0 | 1

9. Primary Outcome: Part 2 Arm 1b: Objective Response Rate (ORR)
Description: as for outcome 7
Time Frame: From start of treatment up to 104 weeks
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2 (mCRPC): Arm 1b: BNT112
Number analyzed (Participants) | 25
percentage of participants | 12.0 [2.5 to 31.2]
Statistical Analysis 1: Comparison: Part 2 (mCRPC): Arm 1b: BNT112; Test type: Superiority; p = 0.0541, Binomial test

ADVERSE EVENTS:
Time Frame: From Baseline up to 30 days after the last dose of BNT112 (for Part 1 and Part 2 Arm 1b and 3) or up to 90 days after the last dose of cemiplimab (for Part 2, Arm 1a and Arm 2) (up to 4 years and 1 month). As per the protocol, non-SAEs with an onset date more than 30 days after the last dose of BNT112 or 90 days after the last dose of cemiplimab (for Part 2, Arm 1a and Arm 2) are only reported below if assessed as related to IMP by the investigator.
Description: Analysis (including all-cause mortality) was performed on safety set. One participant in the Part 1 (mCRPC): BNT112 arm withdrew from the study 13 days after receiving their last dose and is reported in the participant flow section as having withdrawn from the study (based on the ITT population). However, the subject died within 30 days of their last dose so counted in the all-cause mortality for this arm which is based on the safety set.
Arm/Group | Part 1 (mCRPC): BNT112 | Part 2 (mCRPC): Arm 1a: BNT112 + Cemiplimab | Part 2 (mCRPC): Arm 1b: BNT112 | Part 2 (LPC): Arm 2: BNT112 + Cemiplimab | Part 2 (LPC): Arm 3: BNT112
All-Cause Mortality (participants affected / at risk) | 7/9 | 17/28 | 13/27 | 1/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 5/9 | 5/28 | 9/27 | 2/5 | 2/6
Other Adverse Events (participants affected / at risk) | 8/9 | 28/28 | 26/27 | 5/5 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 (mCRPC): BNT112 (N=9) | Part 2 (mCRPC): Arm 1a: BNT112 + Cemiplimab (N=28) | Part 2 (mCRPC): Arm 1b: BNT112 (N=27) | Part 2 (LPC): Arm 2: BNT112 + Cemiplimab (N=5) | Part 2 (LPC): Arm 3: BNT112 (N=6)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Right ventricular failure (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 1 | 0 | 0
Appendicitis perforated (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pelvic abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 2 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Ureteric obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Urethral obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 (mCRPC): BNT112 (N=9) | Part 2 (mCRPC): Arm 1a: BNT112 + Cemiplimab (N=28) | Part 2 (mCRPC): Arm 1b: BNT112 (N=27) | Part 2 (LPC): Arm 2: BNT112 + Cemiplimab (N=5) | Part 2 (LPC): Arm 3: BNT112 (N=6)
Anaemia (Blood and lymphatic system disorders) | 4 | 8 | 4 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 3 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 1 | 0 | 1
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 1
Hypothyroidism (Endocrine disorders) | 0 | 2 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 3 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 2 | 3 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 6 | 0 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 6 | 6 | 1 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 3 | 4 | 0 | 0
Asthenia (General disorders) | 0 | 2 | 2 | 0 | 0
Chest pain (General disorders) | 1 | 1 | 0 | 0 | 0
Chills (General disorders) | 1 | 16 | 6 | 1 | 4
Fatigue (General disorders) | 2 | 10 | 5 | 1 | 2
General physical health deterioration (General disorders) | 0 | 2 | 0 | 0 | 0
Influenza like illness (General disorders) | 2 | 5 | 5 | 3 | 2
Injection site reaction (General disorders) | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 3 | 2 | 1 | 1
Pyrexia (General disorders) | 6 | 17 | 16 | 1 | 2
Cytokine release syndrome (Immune system disorders) | 1 | 0 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 4 | 5 | 0 | 0
Coronavirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 2 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 2 | 0 | 0 | 1
Amylase increased (Investigations) | 0 | 0 | 1 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 3 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 2 | 4 | 1 | 1 | 0
Blood creatinine increased (Investigations) | 2 | 0 | 2 | 1 | 1
Blood pressure increased (Investigations) | 0 | 2 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 1 | 2 | 1 | 0
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 3 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 2 | 3 | 0 | 1 | 0
Lipase increased (Investigations) | 0 | 0 | 1 | 1 | 1
Platelet count decreased (Investigations) | 0 | 2 | 0 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 1 | 0 | 0 | 1
Weight decreased (Investigations) | 2 | 1 | 2 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2 | 2 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 6 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 4 | 3 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 3 | 1 | 1 | 2
Headache (Nervous system disorders) | 1 | 3 | 2 | 2 | 2
Neuropathy peripheral (Nervous system disorders) | 0 | 2 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 3 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 1 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 2
Pyelocaliectasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 0 | 0 | 1 | 2
Hypertension (Vascular disorders) | 4 | 4 | 5 | 1 | 3
Hypotension (Vascular disorders) | 0 | 0 | 3 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of this trial may be published or presented at scientific meetings. If this is foreseen, the investigator agrees to submit all manuscripts or abstracts to the sponsor before submission. This allows the sponsor to protect proprietary information and to provide comments.

DOCUMENTS (2):
  • Study Protocol (2022-02-23): https://cdn.clinicaltrials.gov/large-docs/98/NCT04382898/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-27): https://cdn.clinicaltrials.gov/large-docs/98/NCT04382898/SAP_001.pdf